CLINICAL TRIAL: NCT02417805
Title: Effects of Remote Ischemic Preconditioning in Cutaneous Microcirculation of Different Wounds
Brief Title: Cutaneous Microcirculation After Remote Ischemic Preconditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Kisch, MD, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-266-2
Record Dates: First submitted 2015-03-12; First posted 2015-04-16 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Burn Injury; Acute Wound; Chronic Wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Second-Degree Burn (Experimental): Group A (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Intervention: Remote Ischemic Preconditioning
- Skin Excision (for Skin Graft) (Experimental): Group B (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of TBSA.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Intervention: Remote Ischemic Preconditioning
- Chronic Wound (Experimental): Group C (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Intervention: Remote Ischemic Preconditioning
- Intact Skin (Active Comparator): Group D (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups A-C must be evident.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Intervention: Remote Ischemic Preconditioning

INTERVENTIONS:
Procedure: Intervention: Remote Ischemic Preconditioning — Remote Ischemik Preconditioning is performed using a Blood Pressure Cuff with a pressure slightly above patients' blood pressure on the upper arm.

SUMMARY:
In plastic and reconstructive surgery, treatment strategies of second-degree burns, superficial wounds and chronic wounds aim at reducing infection and improving microcirculation. Although previous studies indicate that remote ischemic preconditioning (RIPC) can accelerate wound healing, only a few studies focused on the elucidation of its mechanisms of action. Therefore, the aim of this study is to evaluate the microcirculatory effects of remote ischemic preconditioning on second-degree burns, superficial and chronic wounds in a human in-vivo setting for the first time.

ELIGIBILITY:
Inclusion Criteria:

Group A (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.

Group B (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of TBSA.

Group C (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.

Group D (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups A-C must be evident. No soft tissue injury must be evident.

Exclusion Criteria:

General exclusion criteria

* below 18 years of age
* wounds requiring artificial respiration, since consent for the study participation is unobtainable

Exclusion Criteria Groups A, B, D:

* peripheral arterial occlusive disease
* vasculitis
* diabetes mellitus
* chronic kidney or liver disease
* cardiac dysfunction
* arterial hypo- or hypertension

Anamnestic exclusion criteria

* ongoing immunosuppressive or chemotherapy treatment
* drug abuse
* systemic skin diseases
* systemic and local cortisone therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Change in microcirculation (composite measure) | Baseline and 1 minute post-dose
  * capillary blood flow [arbitrary units AU]
  * capillary blood velocity [AU]
  * tissue oxygen saturation [%]
  * relative postcapillary venous filling pressure [AU]

SECONDARY OUTCOMES:
Change in microcirculation (areolar measure) | Baseline, while and 1 minute post-dose
  * tissue oxygen saturation [%]
  * tissue hemoglobin index

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany